CLINICAL TRIAL: NCT01411176
Title: Phase III Placebo-controlled Study of NPO-11 in Patients Undergoing Therapeutic Upper Gastrointestinal Endoscopy (Randomized, Double-blind, Parallel-assignment, Placebo-controlled Study)
Brief Title: Phase III Study of NPO-11 in Patients Undergoing Therapeutic Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPO-11-02/C-02
Record Dates: First submitted 2011-08-02; First posted 2011-08-08 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Cancer
Keywords: upper gastrointestinal endoscopy; suspected gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menthol (Active Comparator): 20 ml NPO-11
  Interventions: Drug: Menthol
- Placebo (Placebo Comparator): 20 ml NPO-11(Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menthol — 20 mL NPO-11 in a prefilled plastic syringe
  Arms: Menthol
Drug: Placebo — The placebo is included same additives as active comparator.
  Arms: Placebo

SUMMARY:
Patients with early gastric cancer, who require therapeutic upper gastrointestinal endoscopy, such as endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD), will receive intragastric spraying of NPO-11 or placebo. The superiority of NPO-11 to placebo as anti-peristaltic agent will be verified in a randomized, double-blind, parallel-assignment design based on the proportion of patients with suppressed gastric peristalsis during the procedures. The degree of gastric peristalsis is assessed by an independent committee.

The safety of NPO-11 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and seven days after administration in comparison with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

inpatients or outpatients of either sex who require therapeutic upper gastrointestinal endoscopy (EMR or ESD) and meet the criteria (1)-(4) below will be enrolled in the study. Patients have to provide written informed consent for voluntary participation in the study. The criteria (2) and (3) will be confirmed by the endoscopic observation just before starting the intended treatment.

1. Patients with an early gastric cancer located in the lower third of the stomach, who require therapeutic upper gastrointestinal endoscopy (EMR or ESD) (except for those with an intended treatment by using a scope of <9 mm in diameter)
2. Differentiated -type intramucosal gastric cancer or the suspected lesion, ≤ 2 cm in size, no ulcer finding
3. Patients with a single intended lesion for the treatment
4. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study beforehand. The criteria (3) to (5) will be confirmed by the endoscopic observation just before starting the intended treatment.

1. Patients with a history of surgery to the upper gastrointestinal tract
2. Patients who require emergency endoscopy
3. Patients with severe gastric stenosis or deformation which makes observation of gastric peristalsis difficult
4. Patients who require emergency endoscopic treatment except for the intended lesion
5. Patients with a lesion extended to the pyloric ring
6. Patients with an ongoing cancer treatment (chemotherapy or radiotherapy)
7. Patients with pacemaker
8. Patients with known bleeding tendency or Patients with difficulty of antithrombogenic agents withdrawal
9. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil
10. Patients with contraindications to glucagon
11. Patients with contraindications to benzodiazepines, pethidine hydrochloride, and epinephrine
12. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
13. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
14. Patients otherwise ineligible for participation in the study in the investigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients had no or mild peristalsis during the therapeutic procedures | 60 minutes
  No or mild gastric peristalsis is defined as when patients have no or suppressed gastric peristalsis during the therapeutic procedure. The degree of gastric peristalsis in the time periods is assessed by an independent committee.

SECONDARY OUTCOMES:
Duration of peristalsis-suppressing effect | 60 minutes
Difficulty level of the therapeutic procedure | 60 minutes
One-piece resection rate with tumor-free margin | 60 minutes
Adverse events and adverse drug reactions | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Tokyo, Japan